CLINICAL TRIAL: NCT01814579
Title: Vaginal Cuff Closure Time Using Unidirectional Barbed Suture in Robotic Hysterectomy, a Randomized Controlled Trial
Brief Title: Vaginal Cuff Closure Time Using Unidirectional Barbed Suture in Robotic Hysterectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Tennessee (Other)
Collaborators: Methodist LeBonheur Hospital System (Unknown); The West Clinic (Unknown)
Responsible Party: Principal Investigator, Adam Mabe, Resident Physician, University of Tennessee
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11-01423-FB; 12-14 (Other: Baptist HealthCare IRB)
Record Dates: First submitted 2013-03-16; First posted 2013-03-20 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2013-03

CONDITIONS: Disease (or Disorder); Gynecological
Keywords: vaginal; cuff; robotic; hysterectomy; vloc; v-loc; vicryl; unidirectional; barbed; suture
MeSH Terms: conditions — Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- V-Loc Vaginal Cuff Closure (Experimental): Patients in this arm will receive vaginal cuff closure with unidirectional barbed suture at time of their robotic hysterectomy.
  Interventions: Device: Unidirectional Barbed Suture (V-Loc)
- Vicryl Vaginal Cuff Closure (Active Comparator): Patients enrolled in this arm will have their vaginal cuff closed with polyglactin 910 (Vicryl) at the time of their robotic hysterectomy.
  Interventions: Device: polyglactin 910 (Vicryl)

INTERVENTIONS:
Device: Unidirectional Barbed Suture (V-Loc) — Patients enrolled in the Unidirectional Barbed Suture arm will have their vaginal cuff closed using this device during their robotic hysterectomy.
  Other Names: V-Loc Wound Closure System
  Arms: V-Loc Vaginal Cuff Closure
Device: polyglactin 910 (Vicryl) — Patients in the Smooth Suture arm will have their vaginal cuff closed with this device during their robotic hysterectomy.
  Other Names: Vicryl
  Arms: Vicryl Vaginal Cuff Closure

SUMMARY:
This study is designed to determine if using the V-Loc Wound Closure System expedites operative time in robotic hysterectomy.

DETAILED DESCRIPTION:
Currently both traditional continuous smooth suture and unidirectional barbed suture techniques are standard of care in robotic hysterectomy and the decision of which to use is at the discretion of the surgeon. By using unidirectional barbed suture in which no knot tying is required, wound closure time may be decreased resulting in decreased operative time. This study was created to compare vaginal cuff closure times using these two techniques.

ELIGIBILITY:
Inclusion Criteria:

* Women being scheduled to have a robotic hysterectomy for benign or malignant disease by the West Clinic Gynecology-Oncology Physicians
* Females age 18+

Exclusion Criteria:

* Patients receiving ongoing radiation therapy to the pelvis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-05 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Vaginal Cuff Closure Time | At time of surgery
  Vaginal cuff closure time will be timed at time of robotic hysterectomy.

SECONDARY OUTCOMES:
Vaginal Cuff Dehiscence | Post Operatively (3 months)
  Patients will be evaluated post operatively by physical examination to determine if a vaginal cuff dehiscence has occurred and will be again screened by phone 3 months post operatively.
Vaginal Cuff Evisceration | Post Operatively (3 months)
  Patients will be evaluated post operatively by physical examination to determine if a vaginal cuff evisceration has occurred and will be again screened by phone 3 months post operatively.
Vaginal Cuff Granulation Tissue Formation | Post Operatively (3 months)
  Patients will be evaluated post operatively by physical examination to determine if a vaginal cuff granulation tissue formation has occurred and will be again screened by phone 3 months post operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Tillmanns, MD, Principal Investigator — University of Tennessee, The West Clinic; Adam Mabe, MD, Principal Investigator — University of Tennessee
Locations (2):
- United States (2):
  - Methodist University Hospital, Memphis, Tennessee
  - The West Clinic, Memphis, Tennessee

REFERENCES:
- [Background] Bradshaw AD, Advincula AP. Incidence and characteristics of patients with vaginal cuff dehiscence after robotic procedures. Obstet Gynecol. 2009 Dec;114(6):1372. doi: 10.1097/AOG.0b013e3181c3f60f. No abstract available. PMID 19935045
- [Background] Siedhoff MT, Yunker AC, Steege JF. Decreased incidence of vaginal cuff dehiscence after laparoscopic closure with bidirectional barbed suture. J Minim Invasive Gynecol. 2011 Mar-Apr;18(2):218-23. doi: 10.1016/j.jmig.2011.01.002. PMID 21354068
- [Background] Einarsson JI, Vellinga TT, Twijnstra AR, Chavan NR, Suzuki Y, Greenberg JA. Bidirectional barbed suture: an evaluation of safety and clinical outcomes. JSLS. 2010 Jul-Sep;14(3):381-5. doi: 10.4293/108680810X12924466007566. PMID 21333192
- [Background] Greenberg JA. The use of barbed sutures in obstetrics and gynecology. Rev Obstet Gynecol. 2010 Summer;3(3):82-91. PMID 21364859
- See also: V-Loc Wound Closure Device Device Information — http://www.covidien.com/vloc/pages.aspx